CLINICAL TRIAL: NCT03270007
Title: Research of Intensive Treatment in Hormone Receptor<10% and Human Epidermal Growth Factor Receptor-2 Negative Breast Cancer Patients With Positive Lymph Node Residual Disease After Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tao OUYANG (Other)
Responsible Party: Sponsor-Investigator, Tao OUYANG, Chairman of Breast Center, Peking University
Organization: Peking University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCP19
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Primary Breast Cancer
MeSH Terms: interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Experimental)
  Interventions: Drug: Vinorelbine
- Control (No Intervention)

INTERVENTIONS:
Drug: Vinorelbine — different from primary chemotherapy(containing anthracycline or paclitaxel)
  Other Names: Intensive treatment
  Arms: Chemotherapy

SUMMARY:
This is a phase IV, single-center, prospective, open-label, randomized,controlled study

ELIGIBILITY:
Inclusion Criteria:

* Female patients, 18≦age ≦66 years
* Biopsy proven lymph node positive, estrogen receptor<10%、progesterone receptor <10% and human epidermal growth factor receptor-2 negative primary breast cancer
* Must have completed neo-adjuvant chemotherapy with a standard regimen(containing both anthracycline and paclitaxel)
* Must have undergone surgery to remove the primary tumor by either a mastectomy or enlarged local excision
* Postoperative residual positive lymph nodes
* Adequate recovery from recent surgery
* No history of other malignancies
* No currently uncontrolled diseased or active infection
* Not pregnant or breast feeding, and on appropriate birth control if of child-bearing potential
* Adequate cardiovascular function reserve with a myocardial infarction within the past six month
* without radiotherapy and chemotherapy contraindication
* Adequate hematologic function with:

  1. Absolute neutrophil count (ANC) ≥1500/mm3
  2. Platelets ≥100,000/ mm3
  3. Hemoglobin ≥10 g/dL
* Adequate hepatic and renal function with:

  1. Serum bilirubin ≤1.5×UNL
  2. Alkaline phosphatase and alanine aminotransferase (ALT) ≤2.5 x ULN. (≤5 x ULN is acceptable in the setting of hepatic metastasis)
  3. BUN between 1.7 and 8.3 mmol/L
  4. Cr between 40 and 110 umol/L
* Knowledge of the investigational nature of the study and Ability to give informed consent
* Ability and willingness to comply with study procedures.

Exclusion Criteria:

* Known or suspected distant metastases
* Concurrent malignancy or history of other malignancy
* Uncontrolled diseases(e.g., heart failure, myocardial infarction within 6 months, arrhythmia, unstable diabetes, hypercalcemia) or active infection
* Geographical, social, or psychological problems that would compromise study compliance
* Known or suspected hypersensitivity to vinorelbine

Ages: 18 Years to 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2017-11-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
distant disease-free survival (DDFS) | 5 years after surgery

SECONDARY OUTCOMES:
relapse-free survival（RFS）、overall survival（OS） | 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Xing Wang, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang X, He Y, Li J, Wang T, Fan Z, Ouyang T. Intensive treatment of triple negative breast cancer with residual positive axillary lymph node after neoadjuvant chemotherapy. BMC Womens Health. 2024 Nov 27;24(1):629. doi: 10.1186/s12905-024-03441-0. PMID 39604957